CLINICAL TRIAL: NCT06799091
Title: Effect Of Neuromodulation on Pain and Quality of Life In Patient With Fibromyalgia Syndrome
Brief Title: Effect Of Neuromodulation In Patient With Fibromyalgia Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rowida Abd Elgleel Sayed Abd Elgleel, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Effect of neuromodulation
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Device: Low frequency TENS
- Low fequency TENS (Active Comparator)
  Interventions: Device: Low frequency TENS

INTERVENTIONS:
Device: Low frequency TENS — Low TENS group participated in twelve sessions of electrical stimulation with low frequency (TENS, 10 Hz/200 μs) was applied with self-adhesive electrodes (size 9 × 5 cm,), in the paravertebral ganglionar region (from T1 to L2). The sessions took place at the same time of the day, lasted 30 min, in an acclimatized room (23 °C) and the intensity of the current was delivered at sensory-level intensity, adjusted every 5 min by the sensory threshold, during the 30 min as tolerated by each subject, but without motor contraction or pain reported by the subject.

SUMMARY:
This study was designed to examine the efficacy of Neuromodulation therapy By using transcutanous electric nerve stimulation( TENS) in Patients With FMS and to provide preliminary evidence regarding its effects on pain ,anxiety and QOL by objectively measuring Cortisol level in FMS patients.

DETAILED DESCRIPTION:
Forty female patients with FM ( age : 20- 45 Years ) participated in the study after suing the consent form . Participants were randomly allocated assigned into 2 equal groups ( control group [ G1 ] and low TENS group [G2 ] ) . Group 1 received selected programs of Physiotherapy including Aerobic exercise and placebo low TENS. Group 2 received low frequency TENS (10 Hz).All participants were assessed for cortisol and pain level by using visual analogues scale Also participants were assessed for QOL by FIBROMYALGIA IMPACT QUESTIONNAIRE (FIQR) . treatment was done 3 sessions per weeks for successive 6 weeks pre and post assessment for all valuable were Done.

ELIGIBILITY:
Inclusion Criteria:

women between 20-45 years old, (ii) diagnoses according to the 2016 American College of Rheumatology criteria for fibromyalgia [1]

- Symptoms have been present at a similar level for at least three months (iii) Absence of other disorders that causes similar symptoms: systemic lupus erethromatosis (SLE), rheumatoid arthritis (RA) and Lyme disease based on laboratory investigations (erythrocyte sedimentation rate (ESR), Anti anti-cyclic citrullinated peptide (Anti CCP), antinuclear antibody (ANA) and Rheumatoid factor (RF)).

Exclusion Criteria:

* any medical, neurological, or psychiatric illness, use of strong opioids or other painkillers except paracetamol and/or ibuprofen, benzodiazepine, illicit drug or alcohol use, recent use of cannabis, pregnancy, breast feeding, and the presence of pain syndromes other than FM.

Presence of other autoimmune disorders e.g.: rheumatoid arthritis and systemic lupus erethromatosus

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Cortisol level | Six weeks after begining of intervention
  Changes in pain from baseline to six weeks after begining of intervention

SECONDARY OUTCOMES:
Fibromyalgia impact questionaire | Six weeks after begining of intervention
  Changes of quality of life from baseline to six weeks after begining of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy laps at cairo university, Giza, Egypt